CLINICAL TRIAL: NCT01029431
Title: Evaluation of the Intubating Laryngeal Airway in Children - Phase 2
Brief Title: Evaluation of the Intubating Laryngeal Airway in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Simon Whyte, Principle Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H08-02199
Record Dates: First submitted 2009-12-07; First posted 2009-12-10 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Intubating Laryngeal Airway
Keywords: intubating laryngeal airway; pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects will have both Air-Q ILA & PLMA
  Interventions: Device: AirQ Intubating Laryngeal Airway

INTERVENTIONS:
Device: AirQ Intubating Laryngeal Airway — After induction of anaesthesia in each child, either a PLMA or an Air-Q® ILA of the weight-appropriate size will be inserted & the evaluation described below will be conducted. The first LMA will then be removed & the other device inserted & assessed. The order in which the LMA devices are inserted will be determined using block randomisation, with random block sizes, after recruitment & before induction of anesthesia. The anesthesiologist will insert the LMAs using the manufacturer's recommended technique, & inflate the cuff to the manufacturer's recommended intracuff pressure of 60 cm H2O. Intracuff pressure will be measured with a digital pressure cuff monitor.

SUMMARY:
The Air-Q® intubating laryngeal airway (Air-Q® ILA) is an extraglottic device specifically engineered for use both as a stand-alone laryngeal mask airway (LMA) and as a rescue device or "Plan B" device in the event of a difficult airway. As with some other types of LMA, it is then possible to insert an endotracheal tube (ETT) through the Air-Q® ILA, either blindly or mounted on a fibreoptic bronchoscope (FOB), to achieve endotracheal intubation. The objective of this study is to compare the Air-Q® ILA's performance to the current best option, the PLMA.

DETAILED DESCRIPTION:
Hypothesis: The hypothesis is that, for each of the four ILA size categories, 1.0, 1.5, 2.0 & 2.5:

H0: Mean oropharyngeal leak pressure with Air-Q® ILA= mean oropharyngeal leak pressure with PLMA.

H1: Mean oropharyngeal leak pressure with Air-Q® ILA≠ mean oropharyngeal leak pressure with PLMA.

Background: The laryngeal mask airway (LMA) is used during pediatric anesthesia for routine and difficult airway management. The ideal pediatric LMA device would provide excellent sealing at low pressure; facilitate easy endotracheal intubation; and be available in pediatric sizes. Such a device would be an invaluable addition to difficult pediatric airway management plans and, by increasing the likelihood of quickly and effectively securing the difficult airway, and decreasing the risk of catastrophic hypoxemia, would increase perioperative safety for children. The Air-Q® ILA is a modified LMA device whose features encompass the characteristics of the ideal LMA. Our objective is to determine whether or not this new airway device is an improvement over the current standard of care.

Specific Objectives:

The objective of this study is to compare the Air-Q® ILA's performance to the current best option, the PLMA.

Methods:

Recruitment of subjects: With ethical and institutional review board approval, and with written parental informed consent, we will recruit children undergoing elective surgery. Children with ASA status IV-V, abnormal or contraindicated cervical spine flexion/extension/rotation, contraindication to LMA placement, or requiring emergency surgery will be excluded. All children will undergo intravenous induction of anesthesia, as per our routine institutional practice.

Administration of Air-Q® ILA: In phase 2, either a PLMA or an Air-Q® ILA will be inserted and assessed. The first LMA will then be removed and the other device inserted and assessed. The order of insertion will be determined by block randomization.

Data analysis: In phase 2, we will compare OLP values using paired t- tests. We will conduct appropriate statistical analysis of the data on the other assessment variables, which are all secondary outcome measures. Descriptive data will be presented as mean ± SD, median (range), counts (percentages or proportions) as appropriate.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Key inclusion and exclusion criteria Inclusion:

1. ASA I-III
2. Ideal body weight as determined from weight/height centile curves (>3rd & <97th centiles).
3. Elective surgery
4. Appropriate subject and procedure for airway management by LMA sizes 1, 1.5, 2 or 2.5 (Weight 0-50 kg).

Exclusion Criteria:

1. ASA status IV-V
2. Emergency surgery
3. Abnormal or contraindicated cervical spine flexion/extension/rotation
4. Contraindication to LMA placement
5. Aspiration risk; gastro-oesophageal reflux disease
6. Clinically significant pulmonary disease
7. Coagulopathy
8. Distorted airway anatomy judged likely to compromise LMA placement
9. Allergy to any LMA components.

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2009-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure is the most commonly reported primary outcome measure of LMA performance. If fresh gas destined for the lung alveoli leaks around the LMA, inadequate ventilation may result, leading to respiratory acidosis. | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Simon Whyte, MD, Principal Investigator — University of British Columbia; Stephan Malherbe, MD, Study Director — University of British Columbia; Andrew Morrison, MD, Study Director — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Department of Anesthesia, Vancouver, British Columbia, Canada